CLINICAL TRIAL: NCT01669083
Title: A Phase I Non-Randomized Multi Cohort, Open Label, Bridging Study to Evaluate the Pharmacokinetics, Safety and Tolerability of GSK557296 in Healthy Women Volunteers After Single and Repeat Dosing
Brief Title: Study to Evaluate the Pharmacokinetics, Safety and Tolerability of GSK557296 in Healthy Women Volunteers After Single and Repeat Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116741
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Embryo Transfer
Keywords: Oxytocin Antagonist; Embryo/Blastocyst Implantation
MeSH Terms: interventions — epelsiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: GSK557296 10 mg (Experimental): GSK557296 10 mg single dose on Day 1 followed by repeat dosing (4 times a day) on Days 2-6
  Interventions: Drug: GSK557296 10 mg
- Cohort 2: GSK557296 150 mg (Experimental): GSK557296 150 mg as a single dose on Day 1 followed by repeat nominal dosing of the same dose (either 2, 3 or 4 times a day based on half-life demonstrated in treatment A) on Days 9-13
  Interventions: Drug: GSK557296 150 mg
- Cohort 3 (Experimental): This study had an adaptive design and additional cohorts may be added depending on the PK profiles of Cohort 1 and Cohort 2. Subjects in this optional Cohort 3 will receive GSK557296 (dose to be determined) as a single dose on Day 1 followed by repeat nominal dosing of the same dose (either 2, 3 or 4 times a day based on half-life demonstrated in Cohort 1 and Cohort 2) on Days 2-6
  Interventions: Drug: GSK557296 dose 3
- Cohort 4 (Experimental): This study had an adaptive design and additional cohorts may be added depending on the PK profiles of Cohort 1 and Cohort 1. Subjects in this optional Cohort 4 will receive GSK557296 (dose to be determined) by PK of prior doses, 10-150 mg single dose on Day 1 followed by repeat dosing (either 2, 3 or 4 times a day dependent on half-life demonstrated in prior groups) on Days 2-6
  Interventions: Drug: GSK557296 dose 4

INTERVENTIONS:
Drug: GSK557296 10 mg — 10 mg single oral dose. Each subject will receive 2 tablets of 5 mg GSK557296 four times a day (QID).
  Arms: Cohort 1: GSK557296 10 mg
Drug: GSK557296 150 mg — 150 mg single oral dose. Each subject will receive multiple tablets of 25 mg GSK557296 either 2, 3 or 4 times a day.
  Arms: Cohort 2: GSK557296 150 mg
Drug: GSK557296 dose 3 — Dose to be determined as a single dose tablet based on half-life demonstrated in Cohort 1 and Cohort 2.
  Arms: Cohort 3
Drug: GSK557296 dose 4 — Dose to be determined by PK of prior doses, based on half-life demonstrated in prior cohorts.
  Arms: Cohort 4

SUMMARY:
GSK557296 is being studied in women for the indication of enhanced embryo and or blastocyst implantation in women undergoing IVF treatment. This study will be the first dosing experience with this compound in women. It is important to characterize the pharmacokinetics of GSK557296 in women to determine the most appropriate doses and dosing regimens for future clinical studies. Understanding the pharmacokinetics of GSK557296 in women will also enable more accurate characterization of any exposure-response relationship in future studies.

Two previous studies with GSK557296 were conducted in men with oral doses ranging from 10 milligram (mg) to 200 mg. GSK557296 is being studied in women for the indication of enhanced embryo and or blastocyst implantation in women undergoing IVF treatment. This is a bridging study to characterize the pharmacokinetics of GSK557296 in women to determine the most appropriate doses and dosing regimens for future clinical studies.

This is a non-randomized, open label, adaptive design study in healthy female volunteers. A maximum total of 48 subjects, will participate in different cohorts. Subjects in Cohort 1 will receive 10 mg single dose followed by repeat dose. A one week break will occur to allow for analysis of the PK data, prior to starting the second Cohort. Subjects in Cohort 2 will receive 150 mg single dose followed by repeat dose. Cohort 3 and Cohort 4 were adaptive based on the requirement of additional doses to be studies after PK data will be analyzed from each of the first 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN)
* Single or QTcF < 450 millisecond (msec); or QTc < 480 msec in subjects with Bundle Branch Block
* Healthy as determined by a responsible and experienced physician
* Female between 18 and 45 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of Child-bearing potential and is abstinent or agrees to use contraception methods to sufficiently minimize the risk of pregnancy during the study.
* Body weight >= 50 kilogram (kg) and Body Mass Index (BMI) within the range 19 to 29.9 kg per meter^2 (inclusive)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result at screening or within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* A positive pre-study drug or alcohol screen
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer), exposure to more than four new chemical entities within 12 months prior to the first dosing day Unable to refrain from the use of prescription or non-prescription drugs, with the exception of Oral contraceptives, within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within a 56 day period
* Pregnant females
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08-16 (Actual); Primary Completion 2013-03-09 (Actual); Study Completion 2013-03-09 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters of 20 mg GSK557296 following single and repeat oral dosing | 7 days
  From the plasma concentration-time data, the following PK parameters will be determined: maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve [AUC(0-t) and AUC(0-infinity)], and apparent terminal phase half-life (t1/2). AUC(0-infinity) or AUC(0-τ) and Cmax following single and repeat doses may be used for assessment of dose proportionality.
Composite of PK parameters of 150 mg GSK557296 following single and repeat oral dosing | 14 days
  From the plasma concentration-time data, the following PK parameters will be determined: maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve [AUC(0-t) and AUC(0-infinity)], and apparent terminal phase half-life (t1/2). AUC(0- infinity) or AUC(0-τ) and Cmax following single and repeat doses may be used for assessment of dose proportionality.
Safety and tolerability of GSK557296 following single and repeat dosing | up to 49 days
  Safety and tolerability parameters assessments include adverse events, clinical laboratory, ECG, vital signs, and concurrent medication

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Mahar KM, Stier B, Fries M, McCallum SW. A single- and multiple-dose study to investigate the pharmacokinetics of epelsiban and its metabolite, GSK2395448, in healthy female volunteers. Clin Pharmacol Drug Dev. 2015 Nov;4(6):418-26. doi: 10.1002/cpdd.210. Epub 2015 Aug 26. PMID 27137713
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116741 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116741?search=study&study_ids=116741#rs
- Available data/document: Clinical Study Report: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116741 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register